CLINICAL TRIAL: NCT03617159
Title: Role of Advanced Magnetic Resonance Imaging in Assessment of Pediatric Cerebral Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammad Farghali Ali, Principal investigator, Assiut University
Other Study IDs: MRI in Pediatric Brain stroke
Record Dates: First submitted 2018-07-25; First posted 2018-08-06 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Pediatric Cerebral Stroke; Brain Infarction/Diagnosis
Keywords: magnetic resonance imaging; diffusion weighted imaging
MeSH Terms: conditions — Brain Infarction; Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Diagnostic Modality

SUMMARY:
Stroke can be ischemic, hemorrhagic, or both. Early recognition and treatment of pediatric stroke are critical in optimizing long-term functional outcomes, reducing morbidity and mortality, and preventing recurrent stroke. Neuroimaging plays a vital role in achieving this goal. Neuroimaging is usually the first step in diagnosis, helping discriminate between ischemic/hemorrhagic strokes and also in the identification of underlying potential causes. Multiparametric magnetic resonance imaging (MRI) plays a crucial role in assessing pediatric cerebral stroke including diffusion-weighted imaging (DWI), susceptibility weighted imaging (SWI) and magnetic resonance angiography (MRA).

DETAILED DESCRIPTION:
Stroke is a neurological injury caused by the occlusion or rupture of cerebral blood vessels. Stroke can be ischemic, hemorrhagic, or both. Ischemic stroke is more frequently caused by arterial occlusion, but it may also be caused by venous occlusion of cerebral veins or sinuses. Hemorrhagic stroke is the result of bleeding from a ruptured cerebral artery or from bleeding into the site of an acute ischemic stroke. Stroke is relatively rare in children but can lead to significant morbidity and mortality. Understanding that children with strokes present differently than adults and often present with unique risk factors will optimize outcomes in children. Early recognition and treatment of pediatric stroke are critical in optimizing long-term functional outcomes, reducing morbidity and mortality, and preventing recurrent stroke. Neuroimaging plays a vital role in achieving this goal. Neuroimaging is usually the first step in diagnosis, helping discriminate between ischemic/hemorrhagic strokes and also in the identification of underlying potential causes MRI is a more sensitive test for early detection of an infarction. Magnetic resonance arteriography (MRA) and magnetic resonance venography (MRV) should also be carried out to confirm vessel patency and define the vascular anatomy. MRA will yield further information about blood flow, and MRV will more reliably identify cerebral venous sinus thrombosis. MRI has a high sensitivity and specificity in the first hours after symptom onset with the potential to both characterize the ischemic pathology and to differentiate ischemic from hemorrhagic lesions at least as accurately as computed tomography (CT). Most common imaging protocol used for acute ischemic stroke is an emergent/urgent stroke protocol MRI with MRA. This usually takes approximately 13 min for the MRI sequences and 19 min with MRA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute pathological changes in the central nervous system CNS within 7 days admitted from outpatient, emergency room, or inpatient department
* Confirmed diagnosis of acute stroke by clinical testings performed by a neurologist
* Signed informed consent from the patient

Exclusion Criteria:

* Any person with a pacemaker, metal implant, claustrophobia, or any other contraindication for MR examination
* Any person with epilepsy, brain tumor.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients admitted to the pediatric neurological intensive care unit with cerebral stroke
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
To compare the diagnostic accuracy of advanced MRI sequences versus the conventional sequences in early pediatric cerebral stroke. | Wiithin the first day of stroke
  To compare the diagnostic accuracy of advanced MRI sequences including diffusion-weighted imaging (DWI and susceptibility weighted imaging (SWI) with the conventional MRI sequences including T1 weighted imaging, T2 weighted imaging and fluid attenuating inversion recovery (FLAIR) in assessing pediatric cerebral stroke in assessing early infarction by DWI and presence of blood signal by SWI and comparing these findings with the MR conventional sequences.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Husson B, Rodesch G, Lasjaunias P, Tardieu M, Sebire G. Magnetic resonance angiography in childhood arterial brain infarcts: a comparative study with contrast angiography. Stroke. 2002 May;33(5):1280-5. doi: 10.1161/01.str.0000014504.18199.0d. PMID 11988604
- [Background] Husson B, Lasjaunias P. Radiological approach to disorders of arterial brain vessels associated with childhood arterial stroke-a comparison between MRA and contrast angiography. Pediatr Radiol. 2004 Jan;34(1):10-5. doi: 10.1007/s00247-003-1109-0. Epub 2003 Dec 10. PMID 14669061